CLINICAL TRIAL: NCT05598996
Title: The YourMove Study: Optimizing Individualized and Adaptive mHealth Interventions Via Control Systems Engineering Methods
Acronym: YourMove
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Arizona State University (Other); University of Michigan (Other); National Cancer Institute (NCI) (NIH); Small Steps Labs, LLC (Unknown)
Responsible Party: Principal Investigator, Eric Hekler, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20733; 1R01CA244777-01A1 (NIH)
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Inactivity, Physical; Sedentary Behavior
Keywords: technology; physical activity; resilience; wearable; mobile application; behavior mechanism; behavior; intervention; text message; ecological momentary assessment; reflection; inactivity; exercise; walking; sedentary; Fitbit; smartwatch; notifications; wellness; EMA
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Behavior

STUDY DESIGN:
Intervention Model Description: The study is a 12-month parallel-group randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COT-Based Intervention (Experimental): The COT-based intervention will include the following to improve both steps/day (move more), and improving minutes/week of MVPA (exercise): adaptive daily steps/day goal-setting plus feedback; positive reinforcement (i.e., points, which translate to gift cards), self-monitoring of both steps/day and min/week MVPA; education about MVPA sent via text message in both conditions; planning support for scheduling bouts of MVPA via SMS in both conditions; and motivational messages sent via SMS in both conditions, and the use of a self-experimentation tool (REFLECT), developed based on prior successful pilot efforts, focused on fostering effective self-regulatory capacities of individuals.
  Interventions: Behavioral: COT-Based Intervention
- Control (No Intervention): The non-COT approach was designed to be an equivalent to emerging standard of care options for digital health worksite wellness programs to increase PA (control) for a 12-month study period. Participants assigned to the non-COT-based (control) group will receive the latest Fitbit Versa smartwatch and will download the Fitbit smartphone app. Unlike the intervention group, the daily step goal and the accompanying number of points will be static (10,000 steps/day; 150 points/day, respectively). The goal will be delivered to participants via the standard Fitbit app features and points will be communicated via email. Participants will also receive a weekly PA goal (150 minutes of MVPA/per week) and the same accompanying motivational and informative texts that the intervention group receives. Control participants will not complete the physical activity and exercise reflection and planning exercise (Reflect).

INTERVENTIONS:
Behavioral: COT-Based Intervention — The COT-based approach uses a controller that runs case-by-case dynamical systems simulations modeling based on answers to daily questions rooted in social cognitive theory to produce ambitious but achievable daily adaptive step goal recommendations. The process for the COT-based approach is as follows: Phase 1) 2-week measurement only; Phase 2) open-loop system identification experiment (meant to create individualized dynamical models for each participant); Phase 3) closed-loop experiment to optimize for PA initiation, and Phase 4) closed-loop experiment to optimize for PA maintenance.
  Arms: COT-Based Intervention

SUMMARY:
The purpose of this study is to determine the efficacy of a new digital health tool that uses a phone and smartwatch to encourage physical activity and increase weekly amounts of Moderate to Vigorous Physical Activity (MVPA) over 12 months among adults compared to a digital health intervention that mimics a standard of care corporate wellness program.

DETAILED DESCRIPTION:
Strong evidence indicates physical activity (PA) reduces risk of bladder, breast, colon, endometrium, esophagus, gastric, and renal cancer, and there is moderate evidence for lung cancer. Individuals aged 25+ who are inactive are at high risk of developing a variety of cancers. Unfortunately, only 1/3 of adults meet guidelines for PA; thus, they are an important group to target. In response, the investigators developed JustWalk, a modular adaptive mobile health (mHealth) intervention that makes daily N-of-1 adjustments to support PA for each person. JustWalk can perform N-of-1 adaptation based on our innovative use of control engineering methods, which the investigators call a control optimization trial (COT).

The YourMove study is a 12-month 2-arm randomized control trial (RCT) designed to assess the efficacy of COT methods in 386 adults aged 25+ who are inactive. The investigators will evaluate the differences in minutes/week of moderate-to-vigorous intensity PA (MVPA), measured via accelerometers, among the COT-optimized (intervention) vs. non-COT intervention designed in accordance with standard of care digital corporate wellness to support physical activity (control) groups at 12 months.

The YourMove Study uses a fully integrated system of modalities that include: 1) a popular consumer-level wearable (e.g., Fitbit Versa) and corresponding app (e.g., the Fitbit app); 2) daily process-level analyses done using the Fitbit Versa and ecological momentary assessment (EMA) measures rooted in social cognitive theory (SCT) constructs to promote behavior change; 3) a highly tailored text messaging system encouraging participants to achieve recommended minutes of physical activity: >150 minutes per week of moderate-to-vigorous physical activity (MVPA); and 4) a self-study tool called "Reflect", which is meant to support individuals in self-experimentation to identify strategies that work for them to fit regular MVPA into their lives. The consumer-level devices and app will be used to self-monitor behavior, and their data will be passively acquired in real-time. A variety of self-reported measures asked daily via EMA enables the measurement of psychosocial factors important for the development of a dynamical SCT model and produces ambitious yet achievable step goals that are adaptive to each individual. Algorithms will be used to automatically deliver text messages to support individually tailored goal setting, performance feedback, and goal review in a highly dynamic style that reflects participants' behavioral progress towards achieving a minimum goal of 150 min/week of MVPA.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-80 years old
* Intend to be available for a 12-month intervention
* Willing and able to attend 3 measurement visits over 12-months
* Willing and able to use a smartphone and text messaging
* Willing and able to use the wearable and corresponding app
* Willing and able to walk and engage in moderate-intensity physical activity
* Healthy enough to participate based on the Physical Activity Readiness Questionnaire
* BMI between 18-40 kg/m^2

Exclusion Criteria:

* Psychiatric or medical conditions that prohibit compliance with the study protocol
* Enrolled in or planning to enroll in a physical activity program during the study period
* Those with a mechanical medical implant, such as a pacemaker

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-08-09 (Estimated); Study Completion 2025-08-09 (Estimated)

PRIMARY OUTCOMES:
Change in minutes of moderate-to-vigorous physical activity (MVPA) | Baseline, 12-months
  Measured using a waist-worn tri-axial accelerometer for 7-days

SECONDARY OUTCOMES:
Change in weight | Baseline, 12-months
  Objectively measured weight in kilograms.
Change in Body Mass Index (BMI) | Baseline, 12-months
  Weight and height will be combined to report BMI in kg/m^2.
Change in waist circumference | Baseline, 12-months
  Weight and height will be combined to report BMI in kg/m^2.
Change in waist-to-hip ratio | Baseline, 12 months
  Waist and hip circumference will be combined to report waist-to-hip ratio in cm/cm.
Change in body composition | Baseline, 12 months
  Total body body composition (fat mass, including a rating of visceral adipose tissue, lean mass, and body water) measured with Bioelectric Impedance Analysis (BIA).
Change in basal metabolic rate | Baseline, 12 months
  Measured with Bioelectric Impedance Analysis (BIA).
Change in systolic blood pressure | Baseline, 12 months
  Systolic blood pressure in mmHg.
Change in diastolic blood pressure | Baseline, 12 months
  Diastolic blood pressure in mmHg.
Change in flexibility | Baseline, 12 months
  Sit and reach test.
Change in grip strength | Baseline, 12 months
  Grip strength of the right and left hands in kilograms with a dynamometer.
Physical activity | Through study completion, up to 12 months
  Measured using Fitbit.
Change in physical activity | Baseline, 12 months
  Assessed through self-report using the Global Physical Activity Questionnaire. The questionnaire is comprised of 16 questions related to physical activity in three settings that include activity at work, travel to and from places, and recreational activities, in addition to sedentary behavior. Metabolic Equivalent (MET) values are assigned to time variables according to intensity of activity, moderate or vigorous, reported in each of the settings. MET values are then used to calculate total physical activity.
Sleep | Through study completion, up to 12 months
  Measured using Fitbit.
Resting heart rate | Through study completion, up to 12 months
  Measured using Fitbit.
Sedentary Behavior | Through study completion, up to 12 months
  Measured using Fitbit.
Change in sleep | Baseline, 12 months
  Assessed through self-report using a modified Pittsburg Sleep Quality Index questionnaire. Participants respond to questions related to sleep duration and how often they have difficulty falling asleep and staying awake, do not get enough rest. A higher score indicates more restful sleep.
Change in resting heart rate | Baseline, 12 months
  Measured by research assistant.
Sedentary Behavior | Baseline, 12 months
  Measured using a waist-worn tri-axial accelerometer.
Change in sedentary Behavior | Baseline, 12 months
  Assessed using the Last 7 Day Sedentary Behavior Questionnaire (SIT-Q-7d), which assesses sitting or lying down in five domains (meals, transportation, occupation, non-occupational screen time, and other sedentary time), thus facilitating the calculation of domain-specific and total sedentary time. Frequency within the last 30 days is assessed on a 5-point response scale, ranging from "never or hardly ever" to "always or almost always".
Physical Activity: Change Strategies | Baseline, 12 months
  Physical Activity: Change Strategies survey consists of 15-items that assess how often participants engage in strategies that help them change their physical activity in the past month using a 5-point response scale ranging from "Never" to "Many times".
Physical Activity Neighborhood Environment | Baseline, 12 months
  Physical Activity Neighborhood Environment survey consists of 17-items that assess the environmental factors for walking and bicycling in various neighborhoods. Higher values from the scale indicate greater environmental support for physical activity.
Social Support for Physical Activity | Baseline, 12 months
  Assessed using the Physical Activity and Social Support Scale which consists of 20-items scale based in five forms of social support - companionship, emotional, instrumental, informational, and validation for physical activity. Participants respond to items on a 7-point Likert scale ranging from "never" to "always", or "not applicable". A higher score indicates individuals who are seeking to change exercise behaviors feel a high level of support from friends and family.
Depression | Baseline, 12 months
  Assessed using the Center for Epidemiologic Studies depression scale which consists of 10-items. Participants respond to items related to how they feel and behave on a 5-point response scale ranging from "Rarely or none of the time" to "All of the time". A score equal to or above 10 is considered depressed.
Anxiety | Baseline, 12 months
  Assessed using the short-form of the state scale of the Spielberger State Trait Anxiety Inventory which consists of 6 items. Participants respond to items related to how they feel on a 4-point response scale ranging from "Not at all" to "Very much".
Self-esteem | Baseline, 12 months
  Assessed using the Rosenberg Self-esteem Scale which consists of 10-items. Participants respond to items related to items related to global self-worth on a 4-point Likert scale ranging from "strongly agree" to "strongly disagree". Higher scores indicate higher self-esteem.
Quality of Well-being | Baseline, 12 months
  Assessed using the Quality of Well-being survey, self-administered version which consists of 71 items. Participants respond to items related to health status and overall well-being over the previous 3 days. Scores are translated to quality-adjusted life years.
Change in Gait Speed | Baseline, 12 months
  Measured using the 25-ft walk test
Change lower extremity functional strength | Baseline, 12 months
  Measured using 5x sit-to-stand test which has participants stand up and sit down as quickly as possible 5 times from a straight-backed chair. Only assessed in participants 50 and older.
Change in balance | Baseline, 12 months
  Assessed with feet in three different positions for 20 seconds each position (feet side by side, feet semi-tandem, and feet full-tandem). All balance testing will be measured using BtrackS balance tracking system, a computerized force plate that will provide a more objective and detailed assessment of balance than administrator observation alone, including total sway measured in centimeters. Only assessed in participants 50 and older.
Change in timed-up-and-go (TUG) | Baseline, 12 months
  Participants will be instructed to stand up from a chair, walk around a cone set up 10 feet away, and return to sit in the chair. Only assessed in participants 50 and older.
Change in aerobic fitness | Baseline, 12 months
  Assessed using a sub-maximal graded exercise test. A treadmill walking protocol at a participant-selected speed with elevation increases every 2 minutes will be employed until the participant reaches 85% of age predicted maximal heart rate (220 bpm - age) or volitional fatigue, whichever occurs first.

OTHER OUTCOMES:
Smoking & Marijuana Use | Baseline, 12 months
  Assessed using modified items from the Customary Drinking and Drug Use Record. Participants will respond to 26 items related to their smoking and marijuana use over the past 6 months.
Alcohol Use | Baseline, 12 months
  Assessed using modified items from the Customary Drinking and Drug Use Record. Participants will respond to 10 items related to their alcohol use over the past 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hekler, PhD, Principal Investigator — University of California, San Diego; Daniel Rivera, PhD, Principal Investigator — Arizona State University
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim M, Mansour-Assi S, El Mistiri M, Park J, Banerjee S, Khan O, De La Torre S, Higgins M, Godino J, Patrick K, Nebeker C, Jain S, Klasnja P, E Rivera D, Hekler E. Optimizing and Testing an Individualized and Adaptive Physical Activity Digital Health Intervention: Protocol for a Control Optimization Trial Embedded Within a Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 15;14:e70599. doi: 10.2196/70599. PMID 40815836
- [Derived] Mistiri ME, Khan O, Martin CA, Hekler E, Rivera DE. Data-Driven Mobile Health: System Identification and Hybrid Model Predictive Control to Deliver Personalized Physical Activity Interventions. IEEE Open J Control Syst. 2025;4:83-102. doi: 10.1109/ojcsys.2025.3538263. Epub 2025 Feb 4. PMID 40626117